CLINICAL TRIAL: NCT02083367
Title: Default Mode Network fMRI Maps as a Predictive Index of Hepatic Encephalopathy Outcome
Status: Completed | Type: Observational
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Niral Patel, MD, OSF Healthcare System
Other Study IDs: OSF-14-001
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Hepatic Encephalopathy; Cirrhosis; Nonalcoholic Steatohepatitis; Hepatitis C
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis; Non-alcoholic Fatty Liver Disease; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hepatic Encephalopathy Group: Disease Group
- Control Group: Healthy Group

SUMMARY:
Investigating the impact of hepatic encephalopathy on default mode networks within the brain to provide more clues with understanding the physiology of consciousness and predicting the reversibility of comatose states.

DETAILED DESCRIPTION:
The proposed study will provide better understanding of the patterns of default mode network (DMN) dysfunction in comatose state of hepatic encephalopathy, may help to further define the boundaries of neuronal circuits involve, and will try to assess the prognostic value of fMRI in reversibility of severe metabolic coma.

ELIGIBILITY:
(Hepatic Encephalopathy Group)

Inclusion Criteria:

* Patient or legally acceptable representative must understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local patient privacy regulations.
* Age 18 or older at the time of informed consent.
* Patients with liver cirrhosis attending the gastroenterology department (inpatient or outpatient) with hepatic encephalopathy from various causes of liver failure (i.e. alcoholic, infectious, carcinomatous or toxic).
* The patients will be selected applying Child Pughs score and West Raven classification for hepatic encephalopathy.
* All patients participating in the study will undergo a full neurological exam, 30 min routine EEG recording and neuropsychological evaluation along with the f-MRI study.

(Hepatic Encephalopathy Group)

Exclusion Criteria:

* History of alcohol consumption or illicit drug use within past 3 months.
* Patients with underlying psychiatric or neurologic illness (i.e. schizophrenia, untreated major depressive disorder, epilepsy, neurodegenerative dementia, etc.) resulting in unrelated to encephalopathy impairment of consciousness and/or alteration of normal mental capacity.
* Patients after head injury or with advanced pulmonary, renal, or other than liver failure metabolic disorder (such as severe hypoxia, hypo/hyperglycemia, metabolic acidosis or alkalosis).
* Patients requiring sedation for MRI.
* Pregnant women.

(Normal Control Group)

Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Be age 18 or older at the time of informed consent.
* Subjects must be right handed, be free from any neurological injury, be free from any neurological diseases, be free from any psychological diseases, have a baseline Blood pressure < 140/90, not currently be taking any mind altering medications (including antidepressants, anxiolytics, or opioid/narcotic pain medications), and not have claustrophobia

(Normal Control Group)

Exclusion Criteria:

* Unwillingness or inability to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol.
* History of alcohol consumption 1 week prior to the MRI.
* Illicit drug use within past 3 months.
* Patients requiring sedation for MRI.
* Pregnant women.
* Any other condition, clinical finding, or reason that, in the opinion of the Investigator, is determined to be unsuitable for enrollment into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Hospital Gastroenterology Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Functional MRI imagining | Participants will be followed until all study assessments have been completed, an expected average 4 weeks.
  4 Paradigms:
  1. Resting
  2. Tactile Touch
  3. Motor
  4. Auditory

SECONDARY OUTCOMES:
EEG Testing | Participants will be followed until all study assessments have been completed, an expected average 4 weeks.
Neuropsychological Testing | Participants will be followed until all study assessments have been completed, an expected average 4 weeks.
  WAIS-III PHES Digit Span and Trails
Neurological Examination | Participants will be followed until all study assessments have been completed, an expected average 4 weeks.
Serum Ammonia Level | Participants will be followed until all study assessments have been completed, an expected average 4 weeks.
  Hepatic Encephalopathy Group only

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Bhatia, MD, Principal Investigator — OSF Healthcare System; Hrachya Nersesyan, MD, Principal Investigator — OSF Healthcare System
Locations (1):
- OSF Saint Francis Medical Center, Peoria, Illinois, United States

REFERENCES:
- [Background] Baars BJ. Global workspace theory of consciousness: toward a cognitive neuroscience of human experience. Prog Brain Res. 2005;150:45-53. doi: 10.1016/S0079-6123(05)50004-9. PMID 16186014
- [Background] Bluhm RL, Osuch EA, Lanius RA, Boksman K, Neufeld RW, Theberge J, Williamson P. Default mode network connectivity: effects of age, sex, and analytic approach. Neuroreport. 2008 May 28;19(8):887-91. doi: 10.1097/WNR.0b013e328300ebbf. PMID 18463507
- [Background] Boly M, Phillips C, Tshibanda L, Vanhaudenhuyse A, Schabus M, Dang-Vu TT, Moonen G, Hustinx R, Maquet P, Laureys S. Intrinsic brain activity in altered states of consciousness: how conscious is the default mode of brain function? Ann N Y Acad Sci. 2008;1129:119-29. doi: 10.1196/annals.1417.015. PMID 18591474
- [Background] Boly M, Tshibanda L, Vanhaudenhuyse A, Noirhomme Q, Schnakers C, Ledoux D, Boveroux P, Garweg C, Lambermont B, Phillips C, Luxen A, Moonen G, Bassetti C, Maquet P, Laureys S. Functional connectivity in the default network during resting state is preserved in a vegetative but not in a brain dead patient. Hum Brain Mapp. 2009 Aug;30(8):2393-400. doi: 10.1002/hbm.20672. PMID 19350563
- [Background] Buckner RL, Andrews-Hanna JR, Schacter DL. The brain's default network: anatomy, function, and relevance to disease. Ann N Y Acad Sci. 2008 Mar;1124:1-38. doi: 10.1196/annals.1440.011. PMID 18400922
- [Background] Calhoun VD, Adali T, Pearlson GD, Pekar JJ. A method for making group inferences from functional MRI data using independent component analysis. Hum Brain Mapp. 2001 Nov;14(3):140-51. doi: 10.1002/hbm.1048. PMID 11559959
- [Background] Cauda F, Micon BM, Sacco K, Duca S, D'Agata F, Geminiani G, Canavero S. Disrupted intrinsic functional connectivity in the vegetative state. J Neurol Neurosurg Psychiatry. 2009 Apr;80(4):429-31. doi: 10.1136/jnnp.2007.142349. PMID 19289479
- [Background] Coleman MR, Davis MH, Rodd JM, Robson T, Ali A, Owen AM, Pickard JD. Towards the routine use of brain imaging to aid the clinical diagnosis of disorders of consciousness. Brain. 2009 Sep;132(Pt 9):2541-52. doi: 10.1093/brain/awp183. PMID 19710182
- [Background] 10. Coma. New York: Oxford University Press; 2007.
- [Background] Di H, Boly M, Weng X, Ledoux D, Laureys S. Neuroimaging activation studies in the vegetative state: predictors of recovery? Clin Med (Lond). 2008 Oct;8(5):502-7. doi: 10.7861/clinmedicine.8-5-502. PMID 18975482
- [Background] Garrity AG, Pearlson GD, McKiernan K, Lloyd D, Kiehl KA, Calhoun VD. Aberrant "default mode" functional connectivity in schizophrenia. Am J Psychiatry. 2007 Mar;164(3):450-7. doi: 10.1176/ajp.2007.164.3.450. PMID 17329470
- [Background] Gofton TE, Chouinard PA, Young GB, Bihari F, Nicolle MW, Lee DH, Sharpe MD, Yen YF, Takahashi AM, Mirsattari SM. Functional MRI study of the primary somatosensory cortex in comatose survivors of cardiac arrest. Exp Neurol. 2009 Jun;217(2):320-7. doi: 10.1016/j.expneurol.2009.03.011. Epub 2009 Mar 21. PMID 19306870
- [Background] Greicius MD, Kiviniemi V, Tervonen O, Vainionpaa V, Alahuhta S, Reiss AL, Menon V. Persistent default-mode network connectivity during light sedation. Hum Brain Mapp. 2008 Jul;29(7):839-47. doi: 10.1002/hbm.20537. PMID 18219620
- [Background] Greicius MD, Krasnow B, Reiss AL, Menon V. Functional connectivity in the resting brain: a network analysis of the default mode hypothesis. Proc Natl Acad Sci U S A. 2003 Jan 7;100(1):253-8. doi: 10.1073/pnas.0135058100. Epub 2002 Dec 27. PMID 12506194
- [Background] Greicius M. Resting-state functional connectivity in neuropsychiatric disorders. Curr Opin Neurol. 2008 Aug;21(4):424-30. doi: 10.1097/WCO.0b013e328306f2c5. PMID 18607202
- [Background] Jennett B, Bond M. Assessment of outcome after severe brain damage. Lancet. 1975 Mar 1;1(7905):480-4. doi: 10.1016/s0140-6736(75)92830-5. PMID 46957
- [Background] Jeste DV, Palmer BW, Appelbaum PS, Golshan S, Glorioso D, Dunn LB, Kim K, Meeks T, Kraemer HC. A new brief instrument for assessing decisional capacity for clinical research. Arch Gen Psychiatry. 2007 Aug;64(8):966-74. doi: 10.1001/archpsyc.64.8.966. PMID 17679641
- [Background] Laureys S, Boly M, Maquet P. Tracking the recovery of consciousness from coma. J Clin Invest. 2006 Jul;116(7):1823-5. doi: 10.1172/JCI29172. PMID 16823480
- [Background] Mason MF, Norton MI, Van Horn JD, Wegner DM, Grafton ST, Macrae CN. Wandering minds: the default network and stimulus-independent thought. Science. 2007 Jan 19;315(5810):393-5. doi: 10.1126/science.1131295. PMID 17234951
- [Background] McKiernan KA, D'Angelo BR, Kaufman JN, Binder JR. Interrupting the
- [Background] Nersesyan H, Herman P, Erdogan E, Hyder F, Blumenfeld H. Relative changes in cerebral blood flow and neuronal activity in local microdomains during generalized seizures. J Cereb Blood Flow Metab. 2004 Sep;24(9):1057-68. doi: 10.1097/01.WCB.0000131669.02027.3E. PMID 15356426
- [Background] Norton L, Hutchison RM, Young GB, Lee DH, Sharpe MD, Mirsattari SM. Disruptions of functional connectivity in the default mode network of comatose patients. Neurology. 2012 Jan 17;78(3):175-81. doi: 10.1212/WNL.0b013e31823fcd61. Epub 2012 Jan 4. PMID 22218274
- [Background] Raichle ME, MacLeod AM, Snyder AZ, Powers WJ, Gusnard DA, Shulman GL. A default mode of brain function. Proc Natl Acad Sci U S A. 2001 Jan 16;98(2):676-82. doi: 10.1073/pnas.98.2.676. PMID 11209064
- [Background] Raichle ME, Snyder AZ. A default mode of brain function: a brief history of an evolving idea. Neuroimage. 2007 Oct 1;37(4):1083-90; discussion 1097-9. doi: 10.1016/j.neuroimage.2007.02.041. Epub 2007 Mar 6. PMID 17719799
- [Background] Tshibanda L, Vanhaudenhuyse A, Boly M, Soddu A, Bruno MA, Moonen G, Laureys S, Noirhomme Q. Neuroimaging after coma. Neuroradiology. 2010 Jan;52(1):15-24. doi: 10.1007/s00234-009-0614-8. PMID 19862509
- [Background] Vanhaudenhuyse A, Noirhomme Q, Tshibanda LJ, Bruno MA, Boveroux P, Schnakers C, Soddu A, Perlbarg V, Ledoux D, Brichant JF, Moonen G, Maquet P, Greicius MD, Laureys S, Boly M. Default network connectivity reflects the level of consciousness in non-communicative brain-damaged patients. Brain. 2010 Jan;133(Pt 1):161-71. doi: 10.1093/brain/awp313. Epub 2009 Dec 23. PMID 20034928
- [Background] Vincent JL, Patel GH, Fox MD, Snyder AZ, Baker JT, Van Essen DC, Zempel JM, Snyder LH, Corbetta M, Raichle ME. Intrinsic functional architecture in the anaesthetized monkey brain. Nature. 2007 May 3;447(7140):83-6. doi: 10.1038/nature05758. PMID 17476267
- [Background] 29. Weissenborn, Karin, et al.
- [Background] Wijdicks EF, Hijdra A, Young GB, Bassetti CL, Wiebe S; Quality Standards Subcommittee of the American Academy of Neurology. Practice parameter: prediction of outcome in comatose survivors after cardiopulmonary resuscitation (an evidence-based review) [RETIRED]: report of the Quality Standards Subcommittee of the American Academy of Neurology. Neurology. 2006 Jul 25;67(2):203-10. doi: 10.1212/01.wnl.0000227183.21314.cd. PMID 16864809
- [Background] Young GB. Clinical practice. Neurologic prognosis after cardiac arrest. N Engl J Med. 2009 Aug 6;361(6):605-11. doi: 10.1056/NEJMcp0903466. No abstract available. PMID 19657124